CLINICAL TRIAL: NCT06284928
Title: Exploration of Microbial Patterns in Hypertension: A Cross-Sectional Analysis of Gut Microbiota in Newly Diagnosed Patients (MIPHYP-CROSS Study)
Brief Title: Metagenomic Analysis of Gut Microbiota in Untreated and Uncontrolled Hypertensive Patients
Acronym: HyGut
Status: Completed | Type: Observational
Sponsor: Xinjiang Medical University (Other)
Responsible Party: Principal Investigator, Xiang Xie, Head of Hypertension Department, Clinical Professor, Xinjiang Medical University
Other Study IDs: 20240104-01
Record Dates: First submitted 2024-01-30; First posted 2024-02-29 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Hypertension; Gut Microbiota
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Untreated Hypertension Group: This cohort includes participants who have been newly diagnosed with hypertension and have not received any antihypertensive therapy. They serve as the primary population for exploring gut microbiota characteristics associated with the onset of hypertension.
  Interventions: Other: Fecal Sample Collection
- Uncontrolled Hypertension Group: This cohort includes participants with hypertension who are receiving antihypertensive medication but whose blood pressure remains above target levels. They are enrolled to examine gut microbiota patterns associated with poor blood pressure control despite treatment.
  Interventions: Other: Fecal Sample Collection
- Healthy Control Group: This cohort includes healthy adult participants with normal blood pressure (office BP <130/80 mmHg) and no history of hypertension, cardiovascular, metabolic, or gastrointestinal diseases. They serve as the reference population for comparative analyses of gut microbiota composition and function against both untreated and uncontrolled hypertensive patients.
  Interventions: Other: Fecal Sample Collection

INTERVENTIONS:
Other: Fecal Sample Collection — Non-invasive stool sample collection for gut microbiota metagenomic analysis. No drug or behavioral intervention involved.

SUMMARY:
This observational study aims to explore the relationship between gut microbiota composition and blood pressure regulation in patients with hypertension. A total of 192 participants will be enrolled, including newly diagnosed untreated hypertensive patients, patients with uncontrolled hypertension under medication, and healthy controls. Fecal samples will be collected for metagenomic sequencing to identify microbial taxa and functional pathways associated with blood pressure levels. The findings are expected to reveal characteristic microbial patterns linked to hypertension and provide potential microbial targets for improving antihypertensive therapy.

ELIGIBILITY:
Inclusion Criteria

General Inclusion (applies to all participants)

1. Adults aged 18 years or older.
2. Able and willing to provide a stool sample for gut microbiota analysis.
3. Able to understand and sign written informed consent prior to participation.

Cohort-Specific Inclusion

A. Untreated Hypertension Group (Newly Diagnosed)

1. Newly diagnosed hypertension, defined as: Office blood pressure ≥140/90 mmHg, confirmed by at least two measurements on separate visits; or 24-hour ambulatory BP monitoring (ABPM): mean ≥130/80 mmHg, or daytime ≥135/85 mmHg, or nighttime ≥120/70 mmHg.
2. Never received any antihypertensive medication prior to enrollment.

B. Uncontrolled Hypertension Group (On Medication)

1. Established hypertension, under stable antihypertensive therapy for ≥4 weeks.
2. Blood pressure not at target, defined as: Office BP ≥140/90 mmHg, or 24-hour ABPM mean ≥130/80 mmHg (daytime ≥135/85 mmHg, nighttime ≥120/70 mmHg).
3. No planned medication changes until stool sampling is completed.

C. Healthy Control Groups

1. No history of hypertension or antihypertensive medication use.
2. Office BP <130/80 mmHg (average of 2-3 readings).
3. Free from major chronic or gastrointestinal diseases.

Exclusion Criteria

1. Use of antibiotics, probiotics, or prebiotics within the previous 3 months, or bowel preparation for colonoscopy within 4 weeks.
2. Chronic gastrointestinal diseases (e.g., inflammatory bowel disease, irritable bowel syndrome, celiac disease) or history of major gastrointestinal surgery (including bariatric surgery).
3. Presence of major chronic diseases that may confound gut microbiota or blood pressure regulation, including: Coronary artery disease (CAD) or other significant cardiovascular diseases; Diabetes mellitus (type 1 or type 2); Chronic kidney disease (stage ≥3); Chronic liver disease or hepatic failure; Heart failure (NYHA class III-IV); Active malignancy or history of cancer within the past 5 years.
4. Pregnancy or lactation.
5. Acute infection, acute gastrointestinal symptoms, or hospitalization within the past 4 weeks.
6. Special restrictive diets (e.g., ketogenic, elimination, or medically prescribed weight-loss diets) or alcohol/substance abuse that may alter gut microbiota.
7. Any other condition that, in the investigator's opinion, could interfere with participation, data integrity, or sample quality.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consists of adults aged 18 years or older recruited from the outpatient clinics and health examination centers of the First Affiliated Hospital of Xinjiang Medical University. Participants include three groups: newly diagnosed untreated hypertensive patients, hypertensive patients receiving medication but with uncontrolled blood pressure, and healthy controls without hypertension or major chronic diseases. All participants will provide stool samples for gut microbiota metagenomic analysis and basic clinical data collection.
Sampling Method: Non-Probability Sample
Enrollment: 192 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Gut Microbiota Composition Differences Between Hypertensive and Healthy Individuals | Samples will be collected and analyzed once within the cross-sectional study period .
  Comparative analysis of gut microbiota composition, including bacterial diversity, relative abundance, and taxonomic profiles, between newly diagnosed untreated hypertensive patients and non-hypertensive healthy controls. Metagenomic sequencing will be used to identify microbial taxa and functional pathways associated with blood pressure status.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang, China